CLINICAL TRIAL: NCT01558999
Title: A Clinical Study Evaluating the Safety and Efficacy of SI-614 Ophthalmic Solution in Patients With Dry Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seikagaku Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 614/1121
Record Dates: First submitted 2012-03-18; First posted 2012-03-20 (Estimated); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- High concentration SI-614 (Experimental)
  Interventions: Drug: High concentration SI-614
- Low concentration SI-614 (Experimental)
  Interventions: Drug: Low concentration SI-614
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: High concentration SI-614 — 1 drop in each eye 4 times a day
  Arms: High concentration SI-614
Drug: Low concentration SI-614 — 1 drop in each eye 4 times a day
  Arms: Low concentration SI-614
Drug: Vehicle — 1 drop in each eye 4 times a day
  Arms: Vehicle

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of SI-614 solution compared with placebo solution in treating patients with dry eye

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Have provided written informed consent
* Have dry eye in both eyes

Exclusion Criteria:

* Use of contact lenses
* Have an uncontrolled systemic disease
* Have a history of an uncontrolled psychiatric condition, or substance or alcohol abuse
* Women who is pregnant, nursing or planning a pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-03; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in TFBUT | Day 27
Mean change from baseline in symptom score | Day 21 - 27

CONTACTS AND LOCATIONS:
Locations (1):
- SKK Investigational Site, Andover, Massachusetts, United States